CLINICAL TRIAL: NCT00827372
Title: A Phase II Study of VEGF Inhibition in Patients With Unilateral Upper Extremity Lymphedema Following Treatment for Cancer
Brief Title: A Study of Vascular Endothelial Growth Factor (VEGF) Inhibition in Patients With Unilateral Upper Extremity Lymphedema Following Treatment for Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kathy Miller (Other)
Responsible Party: Sponsor-Investigator, Kathy Miller, Ballvé-Lantero Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0811-15 /IUCRO-0248
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib Treatment (Experimental): Pazopanib 800 mg orally once each day (maximum total duration of treatment = 24 weeks)
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib will be administered at a starting dose of 800 mg orally once each day.
  Other Names: GW786034

SUMMARY:
The major purpose of this study is to determine if a new drug called pazopanib decreases lymphedema in subjects previously treated for cancer. Lymphedema, or swelling of the arm, is a result of damage to the lymphatic vessels in the arm during surgery and/or radiation. The damaged vessels can not adequately drain fluid from the arm, resulting in increased pressure and swelling. Pazopanib has not previously been studied as a treatment for lymphedema.

DETAILED DESCRIPTION:
Pazopanib inhibits the growth of blood vessels in tumors by inhibiting a protein called vascular endothelial growth factor (commonly called VEGF). Pazopanib is not currently approved by the US Food and Drug Administration (FDA) and therefore considered an experimental medication.

High levels of VEGF cause blood vessels to leak fluid, increasing the pressure in tumors similar to the increased pressure in lymphedema. Previous studies have found that treatment with pazopanib decreases the fluid pressure in tumors. That is why we think pazopanib might be an effective treatment for lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Have unilateral lymphedema of the ipsilateral arm attributed to prior surgical treatment or radiation therapy for cancer that is severe enough to warrant therapy in the opinion of the patient and treating physician.
* All patients must have greater than a 3 cm total difference in arm circumference between the affected and unaffected arm measured at five defined points (see protocol).
* Be at least 18 years of age
* Have adequate organ function as specified in the protocol.
* Agree to use effective contraceptive methods during the course of the study if the patient has child-producing potential
* Have an ECOG performance status of 0 or 1

Exclusion Criteria:

* Pregnant, lactating, or unwilling to use appropriate birth control
* Active infection
* Patients may not have clinically significant cardiovascular disease including myocardial infarction within 6 months prior to initiation of therapy, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, grade II or greater peripheral vascular disease, uncontrolled hypertension defined as SBP>160 or DBP>90. Patients may not have any prior history of cerebrovascular disease including TIA or stroke.
* Locally recurrent or metastatic disease
* Concurrent therapeutic anticoagulation or any history of DVT or PE.
* Major surgery within 4 weeks of starting protocol therapy (non-operative biopsy or placement of a vascular access device is not considered major surgery)
* Radiation therapy or chemotherapy within the past 6 weeks or currently undergoing radiation therapy or chemotherapy (Concurrent adjuvant hormonal therapy is allowed.)
* Altered the physical therapy regimen within the past month
* Indwelling venous device in the ipsilateral arm
* Bilateral lymphedema
* Concomitant requirement for medication classified as substrates for the CYP450 enzymes and listed as prohibited in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — IU Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was to enroll 14-15 patients. Due to toxicity and enough patients met the definition of response , this study was halted early, leading to a smaller number of subjects analyzed. There were 10 patients at baseline, 7 patients at Cycle 2, Day 1 and 2 patients who completed the 6 cycles of planned treatment.
Groups:
- Overall Study: All patients who were treated
Period: Overall Study
Arm/Group | Overall Study
Started | 10
Completed | 2
Not Completed | 8
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Volume Ipsilateral Lymphedema in Arm
Description: The primary endpoint will be change in excess arm volume (affected arm volume minus unaffected arm volume) compared to baseline. This will be done at Cycle 2 (29 days) and Cycle 6 (174 days).
Time Frame: Baseline through Cycle 6, Day 1
Population: All patients with non-missing results. There were 10 patients at baseline, 7 patients at Cycle 2, Day 1, and 2 patients who completed the 6 cycles of treatment.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Overall Study
Number analyzed (Participants) | 10
mL
  Change from Baseline to Cycle 2, Day 1 | -161.0 (189.7) [0 to 0]
  Change from Baseline to Cycle 6, Day 1 | -372.8 (233.2)
Statistical Analysis 1: Comparison: Overall Study; With a sample size of 14 evaluable subjects, we will have 80% power to detect a change in excess arm volume of .8 standard deviations using a two-sided paired t-test. We will have 90% power to detect a difference of .9 standard deviations. A Paired T-Test was used to test the difference in arm volume from the second baseline measurement to Cycle 2 only; Test type: Superiority or Other; p = 0.0658, t-test, 2 sided

2. Secondary Outcome: Changes in Interstitial Fluid Pressure (ECF Volume) in the Arm
Description: Interstitial fluid pressure was reported at 24 hours. This is the difference in the last-first reading, affected arm.
  To assess the degree of improvement in arm edema as measured by changes in interstitial fluid pressure (ECF volume using an automated device lymphometer)
Time Frame: First 24 hours after drug was administered
Population: All patients with non-missing results at both baseline and at 24 hours.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Overall: All patients who were treated
Arm/Group | Overall
Number analyzed (Participants) | 7
mm Hg | -0.76 (0.28)
Statistical Analysis 1: Comparison: Overall; A Paired T-Test was used to compare the IFP affected at first versus affected at last reading; Test type: Superiority or Other; p = 0.0061, t-test, 2 sided

3. Secondary Outcome: Change in Impedance or ECF Volume in the Arm
Description: Arm impedance was reported at two baseline readings and for Cycle 2, Day 1.
  To assess the degree of improvement in arm edema as measured by changes in arm impedance (ECF volume using an automated device lymphometer). Data reported is the ratio of the impedance in the affected versus unaffected arm
Time Frame: Baseline, and Cycle 2, Day 1
Population: All patients with non-missing results. This includes 8 patients at the first baseline, 10 patients at the second baseline, and 7 patients at Cycle 2, Day 1.
Measure: Median (Standard Deviation); unit: ratio
Arm/Group | Overall
Number analyzed (Participants) | 10
ratio
  Impedence Baseline 1 | 1.39 (0.34)
  Impedence Baseline 2 | 1.43 (0.31)
  Impedence Cycle 2, Day 1 | 1.46 (0.25)
Statistical Analysis 1: Comparison: Overall; A Paired T-Test was used for the difference in the impedance ratio from the second baseline to cycle 2, day 1; Test type: Superiority or Other; p = 0.0143, t-test, 2 sided

4. Secondary Outcome: Number of Patients With Trt Related Grade 2+ AEs
Description: This is the number of patients who had greater than or equal to Grade 2 Adverse Events related to treatment. This also includes the number of patients who had treatment related Grade 2 or greater Adverse Events that lasted more than 2 weeks (14 days) and excluded events of hypertension (labeled as 'special').
Time Frame: End of Treatment
Population: All treated patients
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 10
participants
  Patients with Trt Related Grade 2+ AEs | 9
  Patients with Trt Related Grade 2+ AEs (special) | 7

5. Secondary Outcome: Clinical Benefit as Assessed by Quality of Life Questionnaire (FACT-B+4 Lymphedema Questions)
Description: The quality of life questionnaire (FACT-B+4 lymphedema questions) was given at various timepoints during the study. The values for the subscales are given for baseline, Cycle 1:Day 1, Cycle 2:Day 1, and Cycle 6:Day 1.
  Physical Well-Being (PWB; sum of 7 items, point range 0-28) Social /Family Well-Being (SWB, sum of 7-items, point range 0-28) Emotional Well-Being (EWB; sum of 6-items, point range 0-24) Functional Well-Being (FWB; sum of 7-items, point range 0-28) Additional Concerns (BCS; sum of 9-items, point range 0-36) Arm subscale (AS; sum of 5-items, point range 0-20) -- This was not collected in Cycle 1 or 2.
  Fact-B+4 score=Sum of PWB, SWB, EWB, FWB, BCS, AS, point range 0-164 Trial Outcome Index=Sum of PWB, FWB, BCS, point range 0-92 Fact-G score=sum of PWB, SWB, EWB, FWB, point range 0-108 Fact-B score=sum of PWB, SWB, EWB, FWB, BCS, point range 0-144 Note: The higher the score, the better the outcome
Time Frame: Baseline through Cycle 6, Day 1
Population: All patients with non-missing results. There were 10 patients at baseline/Cycle 1, Day 1, 7 patients at Cycle 2, Day 1, and 2 patients who completed the 6 cycles of treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Overall
Number analyzed (Participants) | 10
Units on a scale
  Cycle 1, Day 1 Physical Well Being | 25.3 (2.8)
  Cycle 1, Day 1 Social Well Being | 24.9 (2.1)
  Cylce 1, Day 1 Functional Well Being | 22.9 (3.9)
  Cylce 1, Day 1 Emotional Well Being | 21.2 (2.5)
  Cycle 1, Day 1 Additional Concerns | 25.2 (5.5)
  Cycle 1, Day 1 FACT-B+4 Score | 119.5 (11.5)
  Cycle 1, Day 1 Trial Outcome Index | 73.4 (9.2)
  Cycle 1, Day 1 FACT G Score | 94.3 (7.6)
  Cycle 1, Day 1 FACT B Score | 119.5 (11.5)
  Cycle 2, Day 1 Physical Well Being | 22.0 (3.8)
  Cycle 2, Day 1 Social Well Being | 25.8 (2.1)
  Cycle 2, Day 1 Functional Well Being | 21.1 (4.5)
  Cycle 2, Day 1 Emotional Well Being | 20.8 (3.4)
  Cycle 2, Day 1 Additional Concerns | 29.8 (3.7)
  Cycle 2, Day 1 FACT-B+4 Score | 119.6 (11.5)
  Cycle 2, Day 1 Trial Outcome Index | 73.0 (9.1)
  Cycle 2, Day 1 FACT G Score | 89.8 (9.2)
  Cycle 2, Day 1 FACT B Score | 119.6 (11.5)
  Cycle 6, Day 1 Physical Well Being | 24.5 (0.7)
  Cycle 6, Day 1 Social Well Being | 27.4 (0.8)
  Cylce 6, Day 1 Functional Well Being | 25.5 (3.5)
  Cylce 6, Day 1 Emotional Well Being | 23.0 (1.4)
  Cycle 6, Day 1 Additional Concerns | 30.9 (2.4)
  Cycle 6, Day 1 FACT-B+4 Score | 140.9 (20.9)
  Cycle 6, Day 1 Trial Outcome Index | 80.9 (5.2)
  Cycle 6, Day 1 FACT G Score | 100.4 (5.1)
  Cycle 6, Day 1 FACT B Score | 131.4 (7.5)

ADVERSE EVENTS:
Time Frame: Adverse Events are reported from the beginning of study until the end of the study, up to 28 weeks.
Description: There were no serious adverse events entered in this trial.
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=10)
VISION-BLURRED VISION (Eye disorders) | 1 (1)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - ORAL CAVITY (Gastrointestinal disorders) | 5 (5)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 6 (6)
FLATULENCE (Gastrointestinal disorders) | 1 (1)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 4 (4)
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 1 (1)
PAIN - ORAL-GUMS (Gastrointestinal disorders) | 1 (1)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 6 (6)
VOMITING (Gastrointestinal disorders) | 2 (2)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 8 (8)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 2 (2)
SWEATING (DIAPHORESIS) (General disorders) | 1 (1)
ALKALINE PHOSPHATASE (Investigations) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 7 (7)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - NECK NOS (Musculoskeletal and connective tissue disorders) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SKIN (CELLULITIS) (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN - EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN - JOINT (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN - NECK (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN - BACK (Musculoskeletal and connective tissue disorders) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 2 (2)
PAIN - HEAD/HEADACHE (Nervous system disorders) | 1 (1)
PAIN - NEURALGIA/PERIPHERAL NERVE (Nervous system disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 4 (4)
MOOD ALTERATION - DEPRESSION (Psychiatric disorders) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SINUS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 1 (1)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 7 (7)
HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 2 (2)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 3 (3)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 1 (1)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 (3)
RASH: ERYTHEMA MULTIFORME (E.G., STEVENS-JOHNSON SYNDROME, TOXIC EPIDERMAL NECROLYSIS) (Skin and subcutaneous tissue disorders) | 1 (1)
HOT FLASHES/FLUSHES (Vascular disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was to enroll 14-15 patients. Due to toxicity and enough patients met the definition of response, enrollment to this study was halted early, leading to a smaller number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes